CLINICAL TRIAL: NCT01027689
Title: Open-Label, Randomized, Single-Dose, 2-Way Crossover Bioequivalence Study Comparing A New Alprazolam Sublingual Tablet Formulation To A Reference Alprazolam Immediate Release Tablet
Brief Title: Bioequivalence of a New Sublingual and a Reference Alprazolam Immediate Release Tablet Formulation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6131018
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: alprazolam; bioequivalence; sublingual
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alprazolam commercial immediate release oral tablet (Active Comparator)
  Interventions: Drug: alprazolam commercial immediate release oral tablet
- Alprazolam test sublingual tablet (Experimental)
  Interventions: Drug: alprazolam test sublingual tablet

INTERVENTIONS:
Drug: alprazolam commercial immediate release oral tablet — 1 mg tablet, single dose
  Other Names: Xanax
  Arms: Alprazolam commercial immediate release oral tablet
Drug: alprazolam test sublingual tablet — 1 mg tablet, single dose
  Arms: Alprazolam test sublingual tablet

SUMMARY:
This study tests the assumption that the bioavailability of alprazolam from a new sublingual formulation is the same as that from an existing commercial immediate release tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects
* BMI 17.5 - 30.5
* Must provide informed consent

Exclusion Criteria:

* Clinically significant disease
* Narrow angle glaucoma
* Positive drug screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Alprazolam bioavailability assessed as area under the concentration-time curve (AUC) and maximum concentration (Cmax) | 11 days

SECONDARY OUTCOMES:
Alprazolam time of maximum concentration (Tmax) and half life | 11 days
Adverse events, clinical laboratory tests, vital signs | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131018&StudyName=Bioequivalence%20of%20a%20new%20sublingual%20and%20a%20reference%20alprazolam%20immediate%20release%20tablet%20formulation